CLINICAL TRIAL: NCT03787706
Title: Electromyographic Changes in the Cranio-Cervical Flexion Test After Dry Needling of the Upper Trapezius Muscle in Patients With Mechanical Neck Pain
Brief Title: Dry Needling and Electromyographic Changes in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director of Department, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC3010201812618
Record Dates: First submitted 2018-12-22; First posted 2018-12-26 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Neck Pain
Keywords: Neck Pain; Trigger points; Dry needling; Cranio-cervical flexion test
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Patients will receive dry needling over active trigger points in the upper trapezius muscle
  Interventions: Other: Dry Needling
- Manual Therapy (Active Comparator): Patients will receive a manual compression for 30seconds over active trigger points in the upper trapezius muscle
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Dry Needling — Patients will receive dry needling over active trigger points in the upper trapezius muscle
  Arms: Dry needling
Other: Manual Therapy — Patients will receive a manual compression for 30seconds over active trigger points in the upper trapezius muscle
  Arms: Manual Therapy

SUMMARY:
There is evidence suggesting that patients with mechanical neck pain exhibit higher activity of the superficial neck flexor muscles during the execution of the cranio-cervical flexion test. In addition, some studies have reported the presence of active trigger points in the neck flexor and extensor muscles. Since preliminary evidence suggests that trigger points can affect motor control behaviour, it is possible that management of these trigger points with dry needling could be effective for improving muscle activity during low-load activities, such as the cranio-cervical flexion test. Therefore, the aim of this study will be to investigate the effects on electromyographical activity, pressure pain thresholds and cervical range of motion after the application of dry needling over active TrPs in the upper trapezius muscle in patients with mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

Generalized neck-shoulder pain with symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature.

Exclusion Criteria:

* whiplash injury;
* previous cervical or thoracic surgery;
* cervical radiculopathy or myelopathy;
* diagnosis of fibromyalgia syndrome;
* having undergone physical therapy in the previous 6 months;
* less than 18 or greater than 55 years of age
* fear to needles

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in electromyographic activity of the neck superficial flexor muscles before and after the intervention | Baseline and 5 minutes after treatment
  Bipolar surface EMG will be recorded with pairs of electrodes positioned 20mm apart and fixed firmly with an adhesive tape bilaterally over the sternocleidomastoid, the anterior scalene, the upper trapezius and the splenius capitis muscles.

SECONDARY OUTCOMES:
Changes in neck pain intensity with a numerical pain rate scale before and after the intervention | Baseline and 5 minutes after treatment
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to assess spontaneous neck pain intensity
Changes in widespread pressure pain sensitivity before and after the intervention | Baseline and 5 minutes after treatment
  Pressure pain thresholds will be assessed over C5/C6 zygapophyseal joints, second metacarpal, and tibialis anterior muscle
Changes in cervical range of motion before and after the intervention | Baseline and 5 minutes after treatment
  Active cervical range of motion will be assessed with a Cervical Range of Motion (CROM) device in all cervical motions

CONTACTS AND LOCATIONS:
Locations (1):
- Cesar Fernandez-de-Las-Peñas, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Rodriguez-Jimenez J, Ortega-Santiago R, Bonilla-Barba L, Falla D, Fernandez-de-Las-Penas C, Florencio LL. Immediate Effects of Dry Needing or Manual Pressure Release of Upper Trapezius Trigger Points on Muscle Activity During the Craniocervical Flexion Test in People with Chronic Neck Pain: A Randomized Clinical Trial. Pain Med. 2022 Sep 30;23(10):1717-1725. doi: 10.1093/pm/pnac034. PMID 35179608